CLINICAL TRIAL: NCT01137942
Title: Helicobacter Pylori and Gastric Cancer - the Role of Cytokine Polymorphism, Cytokine Expression and Expression of TLR on Persistence of Helicobacter Pylori Infection and Development of Gastric Cancer.
Brief Title: The Role of Cathepsin X in Infection With the Helicobacter Pylori
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Srecko Koren, Institute of microbiology and immunology, Medical faculty Ljubljana, Slovenia
Other Study IDs: IMI2010-1; 1000-05-310123 (Other Grant/Funding Number: Slovenian Research Agency (ARRS))
Record Dates: First submitted 2010-06-02; First posted 2010-06-07 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-03

CONDITIONS: Persistence of Infection With Helicobacter Pylori
Keywords: helicobacter pylori; eradication failure
MeSH Terms: interventions — Clarithromycin; Metronidazole; Proton Pump Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Helicobacter pylori strains from patients are stored at -70oC.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- H. pylori eradication failure: Those who eradicated Helicobacter pylori with appropriate antibiotic therapy and those who did not.
  Interventions: Drug: clarithromycin, metronidazole, proton pump inhibitor

INTERVENTIONS:
Drug: clarithromycin, metronidazole, proton pump inhibitor — appropriate dose of antibiotics and proton pump inhibitor
  Other Names: No other names

SUMMARY:
The immune response to Helicobacter pylori (Hp) importantly determines the pathogenesis of infection as well as the success of antibiotic eradication of the bacteria. The investigators want to demonstrate the importance of cathepsin X (CTSX), a cysteine protease, for the Hp eradication success. The diversity of the innate immune response to H. pylori antigens leading to either successful eradication of the infection or maintenance of chronic inflammation is connected to CTSX. The aim of this study is to determine whether H. pylori suppresses the CTSX expression and cytokine secretion in macrophage cell line THP-1 in the individuals that are not capable of eradicating the infection, opposite to H pylori in patients with successful H pylori eradication . The investigators also investigate the possibility whether strain-dependent differences in H. pylori lipopolysaccharide (LPS) influence the CTSX expression and cytokine secretion.

ELIGIBILITY:
Inclusion Criteria:People with helicobacter gastritis and Helicobacter sensitive to antibiotic therapy but failure of therapy -

Exclusion Criteria:People with helicobacter gastritis who did not eradicate Helicobacter pylori because of primary resistance to antibiotics.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators invited people who had problems with H. pylori(Hp) infection. They were tested for Hp and if positive they were enrolled in the study.All patients were treated with appropriate therapy.3 months after antibiotic therapy, the patients were re-examined. The patients that had a positive test were invited to another re-evaluation.If H. pylori sensitive to all antibiotics tested was isolated, we enrolled the patient in the study-7 patients. The investigators took the patient's first isolate and used it to prepare antigens for the study. All patients in the control group, 7 patients, were successfully cured with first attempt of antimicrobial therapy.Seven months after last patient enrolled, all the participants will be re-evaluated to see if they are still infected with Hp.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Evidence that cathepsin X influences on the eradication of Helicobacter pylori confirmed by lower expression of cathepsin X and cytokines in those patients. that can not eradicate Helicobacter pylori. | 7 months after last participant included in the study
  The investigators assume that vast majority of patients, that have problems with eradication of Helicobater pylori, not caused by primary resistence to antibiotics, can not eradicate helicobacter because of inappropriate immune response. The investigators will measure cathepsin X (CTSX) expression and assume that those patients who have low concentrations of CTSX also have inappropriate immune response seen in low levels of cytokines. To treat such patients, you need to give them different and longer antibiotic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Alojz Ihan, MD, PhD, Study Director — Institute of microbiology and immunology, Ljubljana, Slovenia
Locations (1):
- Abakus Medico, Rogaška Slatina, Slovenia